CLINICAL TRIAL: NCT05735184
Title: Phase 1 Study of Venetoclax/Azacitidine or Venetoclax in Combination With Ziftomenib or Standard Induction Cytarabine/Daunorubicin (7+3) Chemotherapy in Combination With Ziftomenib for the Treatment of Patients With Acute Myeloid Leukemia
Brief Title: A Study to Investigate the Safety and Tolerability of Ziftomenib in Combination With Venetoclax/Azacitidine, Venetoclax, 7+3, or 7+3+Quizartinib in Patients With AML
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kura Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KO-MEN-007
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: Acute Myeloid Leukemia; Mixed Lineage Leukemia Gene Mutation; Refractory AML; AML With Mutated NPM1; Acute Myeloid Leukemia Recurrent; Acute Myeloid Leukemia, in Relapse; NPM1 Mutation; KMT2Ar; Myeloid Sarcoma; Nucleophosmin 1-mutated Acute Myeloid Leukemia
Keywords: Leukemia; Myeloid; AML; Hematological malignancy; KMT2A; NPM1; Menin; Acute Leukemia; Newly diagnosed AML; Untreated AML; venetoclax; cytarabine; daunorubicin; KMT2A-r; NPM1 mutation; Refractory AML; Acute Myeloid Leukemia, in Relapse; quizartinib
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Sarcoma, Myeloid; Leukemia; Hematologic Neoplasms | interventions — venetoclax; Azacitidine; Daunorubicin; Cytarabine; quizartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Dose Escalation: Ziftomenib with Venetoclax and Azacitidine in R/R NPM1-m (A-1) (Experimental): Ziftomenib with Venetoclax and Azacitidine in relapsed/refractory NPM1-m AML patients who have failed at least one prior line of therapy
  Interventions: Drug: Ziftomenib; Drug: Venetoclax; Drug: Azacitidine
- Dose Validation/Expansion: Ziftomenib with Venetoclax and Azacitidine in R/R NPM1-m (A-1) (Experimental): Ziftomenib with Venetoclax and Azacitidine in relapsed/refractory NPM1-m AML patients who have failed at least one prior line of therapy
  Interventions: Drug: Ziftomenib; Drug: Venetoclax; Drug: Azacitidine
- Dose Escalation: Ziftomenib with 7+3 in 1L NPM1-m/FLT3 wildtype (A-2) (Experimental): Ziftomenib with 7+3 in newly diagnosed NPM1-m AML patients who are candidates for intensive chemotherapy and must be FLT3 wildtype or ITD ratio <0.05
  Interventions: Drug: Ziftomenib; Drug: Daunorubicin; Drug: Cytarabine
- Dose Validation/Expansion: Ziftomenib with 7+3 in 1L NPM1-m/FLT3 wildtype (A-2) (Experimental): Ziftomenib with 7+3 in newly diagnosed NPM1-m AML patients who are candidates for intensive chemotherapy and must be FLT3 wildtype or ITD ratio <0.05
  Interventions: Drug: Ziftomenib; Drug: Daunorubicin; Drug: Cytarabine
- Dose Validation/Expansion: Ziftomenib with Venetoclax in R/R NPM1-m (A-3) (Experimental): Ziftomenib with Venetoclax in relapsed/refractory NPM1-m AML patients who have failed at least one prior line of therapy
  Interventions: Drug: Ziftomenib; Drug: Venetoclax
- Dose Validation/Expansion: Ziftomenib with Venetoclax and Azacitidine in 1L NPM1-m (A-4) (Experimental): Ziftomenib with Venetoclax and Azacitidine in newly diagnosed NPM1-m AML patients
  Interventions: Drug: Ziftomenib; Drug: Venetoclax; Drug: Azacitidine
- Dose Escalation: Ziftomenib with Venetoclax and Azacitidine in R/R KMT2A-r (B-1) (Experimental): Ziftomenib with Venetoclax and Azacitidine in relapsed/refractory KMT2A-r AML patients who have failed at least one prior line of therapy
  Interventions: Drug: Ziftomenib; Drug: Venetoclax; Drug: Azacitidine
- Dose Validation/Expansion: Ziftomenib with Venetoclax and Azacitidine in R/R KMT2A-r (B-1) (Experimental): Ziftomenib with Venetoclax and Azacitidine in relapsed/refractory KMT2A-r AML patients who have failed at least one prior line of therapy
  Interventions: Drug: Ziftomenib; Drug: Venetoclax; Drug: Azacitidine
- Dose Escalation: Ziftomenib with 7+3 in 1L KMT2A-r (B-2) (Experimental): Ziftomenib with 7+3 in newly diagnosed KMT2A-r AML patients who are candidates for intensive chemotherapy
  Interventions: Drug: Ziftomenib; Drug: Daunorubicin; Drug: Cytarabine
- Dose Validation/Expansion: Ziftomenib with 7+3 in 1L KMT2A-r (B-2) (Experimental): Ziftomenib with 7+3 in newly diagnosed KMT2A-r AML patients who are candidates for intensive therapy
  Interventions: Drug: Ziftomenib; Drug: Daunorubicin; Drug: Cytarabine
- Dose Validation/Expansion: Ziftomenib with Venetoclax + Azacitidine in 1L KMT2A-r (B-3) (Experimental): Ziftomenib with Venetoclax and Azacitidine in newly diagnosed KMT2A-r AML patients
  Interventions: Drug: Ziftomenib; Drug: Venetoclax; Drug: Azacitidine
- Dose Escalation: Ziftomenib with 7+3+quizartinib in 1L NPM1-m/FLT3-ITD+ AML patients (C-1) (Experimental): Ziftomenib with 7+3 and quizartinib in newly diagnosed NPM1-m and FLT3-ITD+ (with allelic ratio ≥0.05) AML patients who are candidates for IC and eligible to receive FLT3-targeted therapy
  Interventions: Drug: Ziftomenib; Drug: Daunorubicin; Drug: Cytarabine; Drug: Quizartinib
- Dose Validation/Expansion: Ziftomenib with 7+3+quizartinib in 1L NPM1-m/FLT3-ITD+ AML patients (C-1) (Experimental): Ziftomenib with 7+3 and quizartinib in newly diagnosed NPM1-m and FLT3-ITD+ (with allelic ratio ≥0.05) AML patients who are candidates for IC and eligible to receive FLT3-targeted therapy
  Interventions: Drug: Ziftomenib; Drug: Daunorubicin; Drug: Cytarabine; Drug: Quizartinib

INTERVENTIONS:
Drug: Ziftomenib — Oral Administration
  Other Names: KO-539
Drug: Venetoclax — Oral Administration
  Other Names: Venclexta; Venclyxto
  Arms: Dose Escalation: Ziftomenib with Venetoclax and Azacitidine in R/R KMT2A-r (B-1); Dose Escalation: Ziftomenib with Venetoclax and Azacitidine in R/R NPM1-m (A-1); Dose Validation/Expansion: Ziftomenib with Venetoclax + Azacitidine in 1L KMT2A-r (B-3); Dose Validation/Expansion: Ziftomenib with Venetoclax and Azacitidine in 1L NPM1-m (A-4); Dose Validation/Expansion: Ziftomenib with Venetoclax and Azacitidine in R/R KMT2A-r (B-1); Dose Validation/Expansion: Ziftomenib with Venetoclax and Azacitidine in R/R NPM1-m (A-1); Dose Validation/Expansion: Ziftomenib with Venetoclax in R/R NPM1-m (A-3)
Drug: Azacitidine — Subcutaneous or Intravenous Administration
  Other Names: Azadine; Vidaza
  Arms: Dose Escalation: Ziftomenib with Venetoclax and Azacitidine in R/R KMT2A-r (B-1); Dose Escalation: Ziftomenib with Venetoclax and Azacitidine in R/R NPM1-m (A-1); Dose Validation/Expansion: Ziftomenib with Venetoclax + Azacitidine in 1L KMT2A-r (B-3); Dose Validation/Expansion: Ziftomenib with Venetoclax and Azacitidine in 1L NPM1-m (A-4); Dose Validation/Expansion: Ziftomenib with Venetoclax and Azacitidine in R/R KMT2A-r (B-1); Dose Validation/Expansion: Ziftomenib with Venetoclax and Azacitidine in R/R NPM1-m (A-1)
Drug: Daunorubicin — Intravenous Administration
  Other Names: Cerubidine; daunomycin
  Arms: Dose Escalation: Ziftomenib with 7+3 in 1L KMT2A-r (B-2); Dose Escalation: Ziftomenib with 7+3 in 1L NPM1-m/FLT3 wildtype (A-2); Dose Escalation: Ziftomenib with 7+3+quizartinib in 1L NPM1-m/FLT3-ITD+ AML patients (C-1); Dose Validation/Expansion: Ziftomenib with 7+3 in 1L KMT2A-r (B-2); Dose Validation/Expansion: Ziftomenib with 7+3 in 1L NPM1-m/FLT3 wildtype (A-2); Dose Validation/Expansion: Ziftomenib with 7+3+quizartinib in 1L NPM1-m/FLT3-ITD+ AML patients (C-1)
Drug: Cytarabine — Intravenous Administration
  Other Names: cytosine arabinoside (ara-C); Cytosar-U; Tarabine PFS
  Arms: Dose Escalation: Ziftomenib with 7+3 in 1L KMT2A-r (B-2); Dose Escalation: Ziftomenib with 7+3 in 1L NPM1-m/FLT3 wildtype (A-2); Dose Escalation: Ziftomenib with 7+3+quizartinib in 1L NPM1-m/FLT3-ITD+ AML patients (C-1); Dose Validation/Expansion: Ziftomenib with 7+3 in 1L KMT2A-r (B-2); Dose Validation/Expansion: Ziftomenib with 7+3 in 1L NPM1-m/FLT3 wildtype (A-2); Dose Validation/Expansion: Ziftomenib with 7+3+quizartinib in 1L NPM1-m/FLT3-ITD+ AML patients (C-1)
Drug: Quizartinib — Oral Administration
  Other Names: Vanflyta
  Arms: Dose Escalation: Ziftomenib with 7+3+quizartinib in 1L NPM1-m/FLT3-ITD+ AML patients (C-1); Dose Validation/Expansion: Ziftomenib with 7+3+quizartinib in 1L NPM1-m/FLT3-ITD+ AML patients (C-1)

SUMMARY:
Ziftomenib is an investigational drug in development for the treatment of patients with acute myeloid leukemia (AML) with certain genetic alterations.

This protocol has 3 separate arms that will investigate the benefits and risks of adding ziftomenib to standard-of-care (SOC) drug treatments in patients who have AML with certain genetic mutations. Both newly diagnosed and relapsed refractory patients with AML will be assigned to different cohorts based on specific study criteria and physician discretion.

The purpose of this study is to assess the safety, tolerability, and early signs of efficacy of ziftomenib in combination with SOC drugs to treat AML.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients must have a documented NPM1 mutation or KMT2A rearrangement and have either newly diagnosed or relapsed/refractory AML

  * Those intending treatment with intensive chemotherapy in Arm C should be NPM1-m and FLT3-ITD+ with an allelic ratio ≥0.05 and eligible for FLT3-targeted treatment
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Adequate liver, renal, and cardiac function according to protocol defined criteria
* A female of childbearing potential must agree to use adequate contraception as well as a double barrier method from the time of screening through 180 days following the last dose of study intervention. A male of childbearing potential must agree to use abstinence or use a double barrier method of contraception from the time of screening through 180 days following the last dose of study intervention

  * Female patients of childbearing potential who receive quizartinib in Arm C should use a highly effective method of contraception during quizartinib treatment and for 7 months after the last dose

Key Exclusion Criteria:

* Diagnosis of either acute promyelocytic leukemia or blast phase chronic myeloid leukemia
* Known history of BCR-ABL alteration
* Advanced malignant hepatic tumor
* Administration of live attenuated vaccines within 14 days prior to, during, or after treatment until B-cell recovery
* Active central nervous system (CNS) involvement by AML.
* Clinical signs/symptoms of leukostasis or WBC > 25,000 / microliter. Hydroxyurea and/or leukapheresis and/or up to 2 doses of cytarabine if used per institutional SOC for control of leukocytosis are permitted to meet this criterion
* Not recovered to Grade ≤1 (NCI-CTCAE v5.0) from all nonhematological toxicities except for alopecia
* Known clinically active human immunodeficiency virus, active hepatitis B or active hepatitis C infection
* For newly diagnosed cohorts: received prior chemotherapy for leukemia, except hydroxyurea and/or leukapheresis and/or up to 2 doses of cytarabine per institutional standards to control leukocytosis, or prior treatment with all-transretinoic acid for initially suspected acute promyelocytic leukemia
* For relapsed/refractory cohorts: received chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy that is considered to be investigational < 14 days prior to the first dose of ziftomenib or within 5 drug half-lives prior to the first dose of study drug
* Uncontrolled intercurrent illness including, but not limited to, cardiac illness as defined in the protocol
* Mean QT interval corrected for heart rate by Fredericia's formula (QTcF)

  * Arm A and Arm B: >480 ms on triplicate ECGs
  * Arm C: >450 ms on triplicate ECGs
* Uncontrolled infection
* Women who are pregnant or lactating
* An active malignancy and currently receiving chemotherapy for that malignancy or disease that is uncontrolled/progressing
* Patients who have active GVHD requiring >0.5 mg/kg prednisone or any new or increase in immunosuppressants in the prior 2 weeks for GVHD treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2030-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Rate of dose limiting toxicities (DLTs) per dose level (Part 1a only) | During the first 28 days of ziftomenib in combination with SOC backbone treatment (1 cycle)
  Assessed by the NCI-CTCAE v5.0
Descriptive statistics of adverse events | From Cycle 1 Day 1 up to and including 28 days following the end of 36 months of treatment
  Assessed by the NCI-CTCAE v5.0
Complete remission (CR) rate | Until relapse, new anti-cancer therapy, death, or up to 36 months of treatment, whichever occurs first
  Assessed by the ELN 2022 criteria

SECONDARY OUTCOMES:
Composite Complete Remission (CRc) | Until relapse, new anti-cancer therapy, death, or up to 36 months of treatment, whichever occurs first
  Assessed by the ELN 2022 criteria
Morphologic leukemia-free state (MLFS) rate | Until relapse, new anti-cancer therapy, death, or up to 36 months of treatment, whichever comes first
  Assessed by the ELN 2022 criteria
Measurable residual disease (MRD) | Until relapse, new anti-cancer therapy, death, or up to 36 months of treatment, whichever occurs first
  Assessed by multiparameter flow cytometry (MFC) and/or molecular analysis (NGS, PCR)
Median OS | From Cycle 1 Day 1 to date of death from any cause, assessed up to 36 months of treatment
  To assess overall survival of ziftomenib
Proportion of patients alive | From Cycle 1 Day 1 until death from any cause, assessed up to 1 year following start of treatment
  To assess proportion of patients alive at 1 year following start of treatment with ziftomenib
Median EFS | From Cycle 1 Day 1 to treatment failure, hematologic relapse following CR, or death from any cause, whichever comes first, assessed up to 36 months of treatment
  To assess median event free survival
EFS | From Cycle 1 Day 1 to treatment failure, hematologic relapse following CR, or death from any cause, whichever comes first, assessed up to 1 year following start of treatment
  To assess event free survival at 1 year
Median DOR | From time of first remission to relapse or death, whichever occurs first, assessed up to 36 months from start of treatment
  To assess median duration of remission
Proportion of patients who undergo HSCT | From Cycle 1 Day 1 until date of HSCT, assessed up to 36 months of treatment
  To assess proportion of patients who undergo hematopoietic stem cell transplant
TI | From 28 days prior to Cycle 1 Day 1 up to and including 28 days following the end of 36 months of treatment
  To assess rate of transfusion independence
Cmax | Cycle 1; each cycle is 28 days
  Maximum plasma concentration (Cmax) of ziftomenib and metabolites
Tmax | Cycle 1; each cycle is 28 days
  Time to maximum plasma concentration (Tmax) of ziftomenib and metabolites
AUC0-last | Cycle 1; each cycle is 28 days
  Area under the concentration-time curve from time zero to the time of the last quantifiable concentration after dosing (AUC0-last) of ziftomenib and metabolites
AUCtau | Cycle 1; each cycle is 28 days
  Area under the concentration-time curve over a dosing interval (AUCtau) of ziftomenib
Accumulation ratio of ziftomenib and metabolites | Cycle 1; each cycle is 28 days
  To assess accumulation ratio of ziftomenib and metabolites
Cmax of venetoclax | Cycle 1; each cycle is 28 days
  Maximum plasma concentration (Cmax) of venetoclax
Tmax of venetoclax | Cycle 1; each cycle is 28 days
  Time to maximum plasma concentration (Tmax) of venetoclax
AUC0-last of venetoclax | Cycle 1; each cycle is 28 days
  Area under the concentration-time curve from time zero to the time of the last quantifiable concentration after dosing (AUC0-last) of venetoclax
AUCtau of venetoclax | Cycle 1; each cycle is 28 days
  Area under the concentration-time curve over a dosing interval (AUCtau) of venetoclax
Cmax of quizartinib | Cycle 1; each cycle is 28 days
  Maximum plasma concentration (Cmax) of quizartinib
Tmax of quizartinib | Cycle 1; each cycle is 28 days
  Time to maximum plasma concentration (Tmax) of quizartinib
AUC0-last of quizartinib | Cycle 1; each cycle is 28 days
  Area under the concentration-time curve from time zero to the time of the last quantifiable concentration after dosing (AUC0-last) of quizartinib
AUCtau of quizartinib | Cycle 1; each cycle is 28 days
  Area under the concentration-time curve over a dosing interval (AUCtau) of quizartinib

CONTACTS AND LOCATIONS:
Locations (44):
- United States (44):
  - Mayo Clinic - Phoenix, Phoenix, Arizona
  - Moores UC San Diego Cancer Center, La Jolla, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA - Bowyer Oncology Center, Los Angeles, California
  - UC Irvine Health Chao Family Comprehensive Cancer Center, Orange, California
  - University of Colorado, Aurora, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Yale Cancer Center and Smilow Cancer Hospital, New Haven, Connecticut
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Emory Healthcare - The Emory Clinic, Atlanta, Georgia
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - The University of Kansas Medical Center Research Institute, Fairway, Kansas
  - University of Kentucky Markey Cancer Center, Louisville, Kentucky
  - Norton Cancer Institute - St. Matthews, Louisville, Kentucky
  - Ochsner MD Anderson Cancer Center, Jefferson, Louisiana
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - UMass Chan Medical School, Worcester, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers Cancer Institute, New Brunswick, New Jersey
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - New York - Presbyterian / Weill Cornell Medicine, New York, New York
  - Mount Sinai - Ruttenberg Treatment Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Duke Blood Cancer Center, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Cleveland, Ohio
  - The James Cancer Hospital and Solove Research Institute, Columbus, Ohio
  - OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - TriStar Bone Marrow Transplant, Nashville, Tennessee
  - Sarah Cannon Research Institute - St. David's South Austin Medical Center / Texas Oncology South Austin, Austin, Texas
  - UT Southwestern - Simmons Cancer Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No